CLINICAL TRIAL: NCT05753722
Title: An Open-Label Phase 1 Dose-Escalation and Expansion Study Investigating the Safety, Pharmacokinetics, Pharmacodynamics, and Activity of PRTH-101 Alone or in Combination With Pembrolizumab in Adults With Advanced or Metastatic Solid Tumors
Brief Title: A First-in-human Study of PRTH-101 Monotherapy +/- Pembrolizumab in Subjects With Advanced Malignancies
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Incendia Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PRTH-101-0001
Record Dates: First submitted 2023-02-09; First posted 2023-03-03 (Actual); Last update posted 2025-10-31 (Actual); Status verified 2025-09

CONDITIONS: Advanced or Metastatic Solid Tumors; Non Small Cell Lung Cancer; NSCLC
Keywords: Non Small Cell Lung Cancer; NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- PRTH-101 (Experimental): Mono-therapy
  Interventions: Biological: PRTH-101
- PRTH-101 with Pembrolizumab (Experimental): Combo therapy
  Interventions: Biological: PRTH-101; Biological: Pembrolizumab

INTERVENTIONS:
Biological: PRTH-101 — PRTH-101 is a humanized immunoglobulin gamma-1 (IgG1) monoclonal antibody
Biological: Pembrolizumab — PRTH-101 in combination with Pembrolizumab
  Arms: PRTH-101 with Pembrolizumab

SUMMARY:
The goal of this Open-Label Study is to evaluate the safety and tolerability of PRTH-101 alone or in combination with pembrolizumab in adults with advance or metastatic solid tumors.

DETAILED DESCRIPTION:
The goal of this Open-Label Study is to evaluate the safety and tolerability of PRTH-101 alone or in combination with pembrolizumab in adults with advance or metastatic solid tumors.

PRTH-101 is a therapeutic antibody that specifically binds to and blocks DDR1, a protein expressed on tumor cells that binds collagen to make a minimally permeable physical barrier that blocks immune cells from interacting with and attacking tumor cells. These "immune cell-excluded" solid tumors are resistant to attack by the immune system (as well as other existing therapies). By disabling DDR1, the collagen fibers lose alignment and loosen, creating gaps in the tumor barrier, thus allowing T-cells to enter and naturally attack the tumor.

The main question[s] it aims to answer are:

* to evaluate the safety and tolerability of PRTH-101 as mono therapy and in combination with pembrolizumab,
* to determine the recommended Phase 2 dose as mono therapy and in combination with pembrolizumab,
* to evaluate anti-tumor activity of PRTH-101 as mono therapy and in combination with pembrolizumab in selected indications

ELIGIBILITY:
Inclusion Criteria:

1. Subject must be willing and able to read, understand, and sign an Informed Consent Form.
2. Subject must be age ≥18 years.
3. Subject has metastatic or advanced, unresectable malignancy and measurable disease per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 as assessed at Screening, excluding hepatocellular carcinoma, sarcomas, and gliomas.
4. Subject has a pathologically documented advanced/unresectable or metastatic cancer that is refractory to or intolerable to or the subject is unwilling or ineligible to receive standard treatment known to confer benefit or for which no standard treatment is available.
5. Subject must have an Eastern Cooperative Oncology Group performance status (PS) 0-1.
6. Subject must have a predicted life expectancy of ≥3 months.
7. Subject must have the following laboratory values (obtained ≤14 days prior to enrollment):

   1. Calculated creatinine clearance must be ≥30 mL/min by Cockcroft-Gault formula calculation
   2. Total bilirubin ≤1.5 × ULN unless has known history of Gilbert's syndrome (in which case, total bilirubin must be ≤3 × ULN)
   3. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤1.5 × ULN, or ≤3 x ULN in the presence of liver metastases
   4. Hemoglobin ≥9.0 g/dL
   5. Platelets ≥100 × 109 cells/L 9
   6. Absolute neutrophil count ≥1.5 ×10 cells/L (without the use of hematopoietic growth factors)
   7. Corrected QT interval (QTc) ≤470 milliseconds (as calculated by the Fridericia correction formula)
8. Women of child-bearing potential (WOCBP) must have a negative pregnancy test within 3 days prior to first administration of PRTH-101.
9. WOCBP and males with female partners of child-bearing potential must agree to use adequate birth control throughout their participation and for 90 days following the last dose of PRTH-101.
10. Subject must be willing to adhere to the study visit schedule and the prohibitions and restrictions specified in this protocol.
11. Subject must have a site of disease amenable to biopsy and be a candidate for tumor biopsy according to the treating institution's guidelines or have archived tissue available (Section 12.3) at enrollment.

    a. Subjects with sites of disease not amenable to biopsy may be considered after discussion with the Sponsor.
12. The subject is not enrolled in any other clinical trial and is not receiving other therapy directed at their malignancy.
13. The subject is willing to undergo pre-and post-treatment skin biopsies.

Exclusion Criteria:

1. Subject has received prior treatment with systemic agents, including, but not limited to, radio-immunoconjugates, antibody-drug conjugates, immune/cytokines, and monoclonal antibodies (e.g., checkpoint inhibitors) within 28 days or five half-lives of the drug, whichever is shorter.
2. Subject has ongoing toxicity from prior therapy >Grade 1 according to the CTCAE, with the following exceptions. Such exceptions must be assessed by the Investigator (and approved by the Sponsor) as not placing the subject at undue safety risk from participating in this study.

   1. Alopecia, and vitiligo
   2. Grade ≤2 neuropathy
   3. Well-controlled hypo/hyperthyroidism or other endocrinopathies that are well controlled with hormone replacement
3. Subject has undergone a major surgery (excluding minor procedures e.g., placement of vascular access) <2 months prior to administration of PRTH-101.
4. Subject has received radiation therapy <28 days prior to administration of PRTH-101.

   a. Exception: limited (e.g., pain palliation) radiation therapy is allowed prior to and during study treatment as long as there are no acute toxicities, and the subject has measurable disease outside the radiation field.
5. Subject has undergone or is anticipated to undergo organ transplantation including allogeneic or autologous stem-cell transplantation, at any time.
6. Subject has a diagnosis of immunodeficiency, either primary or acquired.
7. Subject has received treatment with systemic steroids or any other form of immunosuppressive therapy within 14 days prior to administration of PRTH-101.

   a. Exception: inhaled or topical (to include mouthwash) steroids and adrenal replacement doses are permitted in the absence of active autoimmune disease.
8. Subject has an active or prior history of autoimmune disease requiring immunosuppressive therapy. Exceptions can be made in discussion with the medical monitor.
9. Subject has a known severe intolerance to or hypersensitivity reactions to monoclonal antibodies, Fc-bearing proteins (e.g., soluble receptors or other Fc fusion proteins), or IV immunoglobulin preparations; prior history of human antihuman antibody response; known allergy to any of the study medications, their analogues, or excipients in the various formulations of any agent.
10. Subject has Central Nervous System (CNS) tumor involvement not definitively treated with surgery or radiation that is active (including evidence of cerebral edema by MRI, or progression from prior imaging study, or has had any requirement for steroids, or clinical symptoms of/from CNS metastases within 28 days prior to study treatment.
11. Subject has leptomeningeal carcinomatosis, regardless of treatment history.
12. Subject has current second malignancy at other sites (exceptions: nonmelanomatous skin cancer, adequately treated in situ carcinoma [e.g., cervical], or indolent prostate cancer under observation). A history of other malignancies is allowed as long as subject has been free of recurrence for ≥2 years, or if the subject has been treated with curative intent within the past 2 years and, in the opinion of the Investigator, is unlikely to have a recurrence.
13. Subject has active and clinically significant bacterial, fungal, or viral infection, including known Hepatitis A, B, or C or HIV (testing not required).
14. Subject has received live vaccines within the past 30 days (inactivated vaccines are allowed; seasonal vaccines should be up to date >30 days prior to administration of PRTH-101).
15. Women who are pregnant or breastfeeding.
16. History of any of the following ≤6 months before first dose:

    a. Congestive heart failure New York Heart Association Grade III or IV b. Unstable angina c. Myocardial infarction d. Unstable symptomatic ischemic heart disease e. Uncontrolled hypertension despite appropriate medical therapy f. Ongoing symptomatic cardiac arrhythmias of > Grade 2 g. Symptomatic cerebrovascular events, or any other serious cardiac condition (e.g., pericardial effusion or restrictive cardiomyopathy); chronic atrial fibrillation on stable anticoagulant therapy is allowed.
17. Subject has any contraindications to the imaging assessments or other study procedures that subjects will be undergoing.
18. Subject has any medical or social condition that, in the opinion of the Investigator, might place a subject at increased risk, affect compliance, or confound safety or other clinical study data interpretation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Estimated)
Dates: Start 2023-03-03 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Evaluate the Adverse Events (AEs), including Serious Adverse Events (SAEs), that occur in patients treated with PRTH-101 | Up to 4 years
  To evaluate the safety of PRTH-101 as assessed by Adverse Events (AEs), including Serious Adverse Events (SAEs) and Dose Limiting Toxicities (DLTs)
Maximum Tolerated Dose | Up to 4 years
  Maximum dose level not requiring dose de-escalation under Bayesian design rules
Pharmacokinetic (PK) profile of PRTH-101 alone and in combination with pembrolizumab | Up to 4 years
  PK parameters for Phase 1a and Phase 1b will include the accumulation ratio.
Pharmacokinetic (PK) profile of PRTH-101 alone and in combination with pembrolizumab | Up to 4 years
  PK parameters for Phase 1a and Phase 1b will include PK maximum concentration (Cmax)
Pharmacokinetic (PK) profile of PRTH-101 alone and in combination with pembrolizumab | Up to 4 years
  PK parameters for Phase 1a and Phase 1b will include observed serum concentration (Tmax)
Pharmacokinetic (PK) profile of PRTH-101 alone and in combination with pembrolizumab | Up to 4 years
  PK parameters for Phase 1a and Phase 1b will include last measurable concentration (Clast),
Pharmacokinetic (PK) profile of PRTH-101 alone and in combination with pembrolizumab | Up to 4 years
  PK parameters for Phase 1a and Phase 1b will include time of last measurable concentration (Tlast,)
Pharmacokinetic (PK) profile of PRTH-101 alone and in combination with pembrolizumab | Up to 4 years
  PK parameters for Phase 1a and Phase 1b will include area under curve up to the last measurable concentration (AUClast)
Pharmacokinetic (PK) profile of PRTH-101 alone and in combination with pembrolizumab | Up to 4 years
  PK parameters for Phase 1a and Phase 1b will include, volume of distribution (Vd,)
Pharmacokinetic (PK) profile of PRTH-101 alone and in combination with pembrolizumab | Up to 4 years
  PK parameters for Phase 1a and Phase 1b will include drug clearance (CL,)
Pharmacokinetic (PK) profile of PRTH-101 alone and in combination with pembrolizumab | Up to 4 years
  PK parameters for Phase 1a and Phase 1b will include the time required for plasma concentration of a drug to decrease by 50% (t1⁄2.)
Anti-tumor activity of PRTH-101 alone and in combination with pembrolizumab | Up to 4 years
  Best overall response as assessed by iRECIST in 1c

SECONDARY OUTCOMES:
To evaluate the incidence and persistence of anti-PRTH-101 antibody formation and its impact on the PK profile of PRTH-101 | Up to 4 years
  Evaluate anti-drug antibody in serum over multiple timepoints and its impact on the PK profile of PRTH-101
To evaluate the incidence and persistence of anti- PRTH-101 antibody formation and its impact on the PK profile of PRTH-101 in combination with pembrolizumab antibody therapy | Up to 4 years
  Evaluate anti-drug antibody in serum over multiple timepoints and its impact on the PK profile of PRTH-101 in combination with pembrolizumab antibody therapy
To evaluate the PK of pembrolizumab | Up to 4 years
  PK parameters for Phase 1b will include the accumulation ratio
To evaluate the PK of pembrolizumab | Up to 4 years
  PK parameters for Phase 1b will include PK maximum concentration (Cmax)
To evaluate the PK of pembrolizumab | Up to 4 years
  PK parameters for Phase 1b will include observed serum concentration (Tmax)
To evaluate the PK of pembrolizumab | Up to 4 years
  PK parameters for Phase 1b will include last measurable concentration (Clast)
To evaluate the PK of pembrolizumab | Up to 4 years
  PK parameters for Phase 1b will include time of last measurable concentration (Tlast)
To evaluate the PK of pembrolizumab | Up to 4 years
  PK parameters for Phase 1b will include area under curve up to the last measurable concentration (AUClast)
To evaluate the PK of pembrolizumab | Up to 4 years
  PK parameters for Phase 1b will include volume of distribution (Vd)
To evaluate the PK of pembrolizumab | Up to 4 years
  PK parameters for Phase 1b will include drug clearance (CL)
To evaluate the PK of pembrolizumab | Up to 4 years
  PK parameters for Phase 1b will include the time required for plasma concentration of a drug to decrease by 50% (t1⁄2.)
To define the PK profile of PRTH-101 together with pembrolizumab | Up to 4 years
  PK parameters for Phase 1b will include accumulation ratio
To define the PK profile of PRTH-101 together with pembrolizumab | Up to 4 years
  PK parameters for Phase 1b will include PK maximum concentration (Cmax)
To define the PK profile of PRTH-101 together with pembrolizumab | Up to 4 years
  PK parameters for Phase 1b will include observed serum concentration (Tmax)
To define the PK profile of PRTH-101 together with pembrolizumab | Up to 4 years
  PK parameters for Phase 1b will include last measurable concentration (Clast)
To define the PK profile of PRTH-101 together with pembrolizumab | Up to 4 years
  PK parameters for Phase 1b will include time of last measurable concentration (Tlast)
To define the PK profile of PRTH-101 together with pembrolizumab | Up to 4 years
  PK parameters for Phase 1b will include area under curve up to the last measurable concentration (AUClast)
To define the PK profile of PRTH-101 together with pembrolizumab | Up to 4 years
  PK parameters for Phase 1b as well as Phase 1c will include volume of distribution (Vd)
To define the PK profile of PRTH-101 together with pembrolizumab | Up to 4 years
  PK parameters for Phase 1b will include drug clearance (CL)
To define the PK profile of PRTH-101 together with pembrolizumab | Up to 4 years
  PK parameters for Phase 1b will include the time required for plasma concentration of a drug to decrease by 50% (t1⁄2.)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Paul Eder, MD, Study Chair — Incendia Therapeutics
Locations (9):
- United States (9):
  - Yale Cancer Center, New Haven, Connecticut
  - Mass General Cancer Center, Boston, Massachusetts
  - Providence Cancer Institute Franz Clinic, Portland, Oregon
  - University of Pittsburgh Medical Center Hillman Cancer Center, Pittsburgh, Pennsylvania
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - Next Oncology, Irving, Texas
  - NEXT Oncology, San Antonio, Texas
  - Next Oncology, Fairfax, Virginia

IPD SHARING:
Plan to Share IPD: No